CLINICAL TRIAL: NCT07047443
Title: Dose Exploration Study of SHR-1811 Combined With Carboplatin in the Treatment of Advanced Breast Cancer With HER2 Expression
Brief Title: SHR-1811 Combined With Carboplatin in the Treatment of Advanced Breast Cancer With HER2 Expression
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Anhui Provincial Cancer Hospital (Other)
Responsible Party: Principal Investigator, Yue-Yin Pan, Chief Physician, Anhui Provincial Cancer Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Anhui1811Carbo
Record Dates: First submitted 2025-06-23; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-A1811 4.8mg/kg + Carboplatin (Experimental): This study adopts the dose escalation pattern of 3+3. Patients with advanced breast cancer expressing HER2 received SHR-A1811 + carboplatin treatment. The dose of SHR-A1811 was fixed at 4.8mg/kg, Q3W, and the initial dose of carboplatin was AUC 2, Q3W. The first cycle of medication (21 days) was used as the tolerance observation period.
  If the subjects cannot tolerate the initial dose combination (intolerance refers to an incidence of DLT ≥33%), the study will be terminated. If it can be tolerated (tolerance refers to the incidence of DLT < 33%), the dose of carboplatin will be increased to AUC 3; If still tolerable, continue to increase the dose of carboplatin to AUC 4.
  Interventions: Drug: SHR- A1811

INTERVENTIONS:
Drug: SHR- A1811 — HER2 ADC

SUMMARY:
To find the optimal dose of carboplatin combined with SHR-A1811 in her2-expressed metastatic breast cancer

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18 to 75 (inclusive of both values).
2. Unresectable or metastatic breast cancer with HER2 positive (IHC 3+ or IHC 2+/ISH+), low HER2 expression (IHC 1+ or IHC 2+/ISH-), or ultra-low HER2 expression (IHC 0 with membrane staining) confirmed by histology or cytology.
3. Failure of standard treatment in the advanced stage.
4. For HER2+ metastatic breast cancer, one can have received second-generation ADC (such as T-DM1) treatment, but cannot have received third-generation ADC (such as T-DXd) treatment. For HER2 low expression or HER2 ultra-low expression metastatic breast cancer, it is necessary to meet the requirement that no ADC drug treatment has been received.
5. For HER2-positive metastatic breast cancer, at the metastatic stage, ≥1 line of anti-HER2 treatment must have been received; For HR-positive metastatic breast cancer with low or ultra-low expression of HER2, it is necessary to meet the failure of CDK4/6 inhibitor treatment at the metastatic stage. For HR-negative metastatic breast cancer with low or ultra-low expression of HER2, it is necessary to have received ≥ first-line chemotherapy at the metastatic stage.
6. The ECOG score is 0 or 1.
7. There is at least one lesion (including measurable or unmeasurable) according to the RECIST v1.1 standard.
8. Adequate organ function.
9. Participants with fertility or their spouses must agree to use appropriate contraceptive measures from the start of the first dose of the study treatment until 120 days after the last dose of the study treatment.
10. Voluntarily join this study and sign the informed consent form.

Exclusion Criteria:

1. Have had other malignant tumors within the past 5 years, excluding cured basal cell carcinoma of the skin and carcinoma in situ of the cervix.
2. There is effusion in the third space that cannot be controlled by methods such as drainage (such as a large amount of ascites, pleural effusion, and pericardial effusion).
3. Clinical researchers who have received surgical treatment (referring to major surgeries for cancer), radiotherapy, chemotherapy, immunotherapy, molecular targeted therapy, biological therapy or other drugs within 4 weeks before the first medication; Those who have received endocrine therapy within two weeks before the first medication.
4. Patients with HER2+ metastatic breast cancer have received treatment with third-generation ADCs (such as T-DXd); Patients with HER2 low-expression or ultra-low-expression metastatic breast cancer who have received any ADC drug treatment.
5. The patient has any active autoimmune diseases or a history of autoimmune diseases that may recur [including but not limited to: autoimmune hepatitis, uveitis, enteritis, pituitinitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism (subjects that can be controlled only through hormone replacement therapy can be included)]; Subjects with skin diseases that do not require systemic treatment, such as vitiligo, psoriasis, alopecia, controlled type 1 diabetes treated with insulin, or asthma that has been completely relieved in childhood and does not require any intervention in adulthood can be included. Asthma patients who require medical intervention with bronchodilators cannot be included.
6. Have a history of immunodeficiency, including a positive HIV test, other acquired or congenital immunodeficiency diseases, or a history of organ transplantation.
7. There are clinically significant cardiovascular diseases, such as severe/unstable angina pectoris, symptomatic congestive heart failure (NYHA ≥ grade II), clinically significant supraventricular or ventricular arrhythmias that require treatment or intervention, and myocardial infarction that occurred within 6 months before the first medication.
8. Subjects with known or suspected interstitial pneumonia; There are other moderate to severe pulmonary diseases that may interfere with drug-related pulmonary toxicity testing or management and seriously affect respiratory function within three months before the first administration, including but not limited to idiopathic pulmonary fibrosis, organized pneumonia/oblusive bronchiolitis, pulmonary embolism, severe asthma, severe chronic obstructive pulmonary disease (COPD), obstructive/restrictive lung disease, etc. And any autoimmune, connective tissue or inflammatory diseases involving the lungs, such as rheumatoid arthritis, Sjogren's syndrome, sarcoidosis, etc., or those who have undergone total lung resection surgery in the past. Subjects who had experienced grade ≥3 interstitial pneumonia during previous treatment with immune checkpoint inhibitors were not allowed to be enrolled in this study.
9. Known hereditary or acquired bleeding predisposition (such as hemophilia, coagulation dysfunction, etc.).
10. There are active hepatitis B (HBsAg positive and HBV DNA≥500 IU/mL), hepatitis C (hepatitis C antibody positive and HCV RNA higher than the upper limit of the normal range), and liver cirrhosis; Or severely infected individuals who need to be controlled with antibiotics, antiviral drugs or antifungal drugs.
11. According to the NCI-CTCAE v5.0 classification, those whose toxicity caused by previous anti-tumor treatment has not yet recovered to grade ≤ Ⅰ (except for alopecia; According to the judgment of the researchers, after consultation with the sponsor, some tolerable chronic grade II toxicities may be excluded.
12. Known allergy to any of the investigational drugs or any of its excipients.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Cancer Hospital, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No